CLINICAL TRIAL: NCT01472770
Title: A Phase II Study of Gemcitabine and Capecitabine for Treatment Resistant, Metastatic Colorectal Cancer
Acronym: GemCaP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GemCap
Record Dates: First submitted 2011-11-01; First posted 2011-11-16 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; Metastatic; Treatment resistant
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine + Capecitabine — Gemcitabine: 1000 mg/m2 intravenously over 30 min. on day 1 in 2-weeks cycles. Capecitabine: Peroral tablet 2000 mg/m2 daily on days 1-7 in 2-weeks cycles.

SUMMARY:
The present study aims to investigate the efficacy and safety of the combination of capecitabine and gemcitabine in heavily pre-treated, treatment resistant metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified colorectal adenocarcinomas
* Age > 18 years
* Metastatic colorectal cancer refractory to 5-FU, oxaliplatin, irinotecan and relevant biological agents.
* Measurable disease according to RECIST 1.1
* ECOG performance status 0, 1 or 2
* Adequate renal, hepatic and haematological function
* Consent to blood samples and available paraffin embedded tumour material for translational research studies
* Fertile males and females (<2 years after last period for women) must use effective birth control.
* Signed Informed consent

Exclusion Criteria:

* Clinically significant concurrent disease.
* Other malignant diseases within 5 years of inclusion in the study, except squamous cell carcinoma of the skin and cervical carcinoma-in-situ.
* Other experimental therapy within 30 days of treatment initiation.
* Patients who are breast feeding, childbearing or of childbearing potential without using dual effective contraception.
* Clinical or radiological evidence of CNS metastasis.
* Planned radiation therapy against target-lesions.
* Known allergy to 5FU/capecitabine or gemcitabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Rate of patients progression free at 3 months | 3 months after start of treatment

SECONDARY OUTCOMES:
Progression free survival | Every 12 weeks
Overall survival | Every 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark